CLINICAL TRIAL: NCT02300909
Title: A Randomized, Single Blind, Controlled Trial of Clinical Outcomes of Dehydrated Human Amnion/Chorion Membrane (dHACM) in Lumbar Decompression and Microdiscectomy Surgery
Brief Title: dHACM in Lumbar Decompression and Microdiscectomy Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MiMedx Group, Inc. (Industry)
Collaborators: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AFLUD001; NCT02380456 (obsolete NCT alias)
Record Dates: First submitted 2014-11-18; First posted 2014-11-25 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Scarring; Spinal Stenosis; Herniated Disc
MeSH Terms: conditions — Cicatrix; Spinal Stenosis; Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dHACM (Experimental): Lumbar Decompression Surgery or Microdiscectomy Surgery with Application of Dehydrated Human Amnion/Chorion Membrane (dHACM)
  Interventions: Procedure: Lumbar Decompression Surgery; Procedure: Microdiscectomy Surgery; Other: Dehydrated Human Amnion/Chorion Membrane (dHACM)
- Surgery without dHACM (Other): Control Group - Lumbar Decompression Surgery or Microdiscectomy Surgery without application of dHACM
  Interventions: Procedure: Lumbar Decompression Surgery; Procedure: Microdiscectomy Surgery

INTERVENTIONS:
Procedure: Lumbar Decompression Surgery — Lumbar Decompression Surgery
Procedure: Microdiscectomy Surgery — Microdiscectomy Surgery
Other: Dehydrated Human Amnion/Chorion Membrane (dHACM) — Application of Dehydrated Human Amnion/Chorion Membrane (dHACM)
  Arms: dHACM

SUMMARY:
Prospective evaluation of the safety and efficacy of dHACM on clinical outcomes in lumbar laminectomy and microdiscectomy patients as assessed by Oswestry Disability Index.

DETAILED DESCRIPTION:
The objective of this prospective study is to evaluate the safety and efficacy of dHACM on clinical outcomes in lumbar laminectomy and microdiscectomy patients randomized to one of two groups: 1) without dHACM (control) or 2) dHACM.

ELIGIBILITY:
Inclusion Criteria:

1. Are 18 (eighteen) years of age or older at the time of surgery.
2. Patients with single- or multi-level spinal stenosis undergoing open lumbar laminectomy, or patients with single-level herniated nucleus pulposus undergoing single-level lumbar microdiscectomy
3. Are willing and able to return for the scheduled follow-up visits, follow post operative instructions and undergo the required radiographic exams for up to 5 time points between 4 weeks and 24 months post-surgery (6 weeks ± 2 weeks, 12 weeks ± 2 weeks, 6 months ±1 month, 1 year±2 months, and 2 years ±2 months post-surgery), including one study MRI-scan at 12 weeks ±2 weeks for the first 20 patients enrolled.
4. Are willing and able to sign study specific informed consent.

Exclusion Criteria:

1. Non-English speaking patients
2. Non-surgical candidate defined as any patient deemed by the surgeon not to be a surgical candidate cannot participate for the following reasons: that patient does not meet indications for lumbar laminectomy or microdiscectomy surgery, patient has a contraindication to surgery such as medical comorbidities, pregnancy, etc.
3. Allergic to aminoglycoside antibiotics
4. Is a prisoner
5. Is involved in worker's compensation or other litigation relative to the spine injury
6. Has a history of drug or alcohol abuse within the last 12 months
7. Is currently participating in another drug or device clinical trial
8. Previous spinal surgery
9. History of deformity, mechanical instability, or spinal fusion requirement
10. History of hard- or soft-tissue spinal infection
11. Has signs or symptoms of any disease, such as autoimmune disease, which could result in allograft failure, or has experienced allograft failure in the past
12. Patients unable to undergo a MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2014-11; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index | 2 years
  Patient Functional Outcomes Questionnaire

SECONDARY OUTCOMES:
Re-operation (Number of patients having re-operation during study) | 2 years
  Number of patients having re-operation during study
Scar formation in revision cases | 2 years
  Dissection of scar formation required at re-operation
Quality of Life (VAS Pain) | 2 years
  VAS Pain
Quality of Life (SF-36) | 2 years
  SF-36
Quality of Life | 2 years
  HSS Lumbar Expectations Survey

OTHER OUTCOMES:
MRI findings in first 20 patients | 3 months post-op

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Hughes, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States